CLINICAL TRIAL: NCT07273292
Title: Autonomic Dysfunction in Neuromyelitis Optica Spectrum Disorder and Multiple Sclerosis : A Comparative Study
Acronym: English Title
Status: Not yet recruiting | Type: Observational
Sponsor: Mohamed Moshref abd alsattar (Other)
Responsible Party: Sponsor-Investigator, Mohamed Moshref abd alsattar, Resident doctor at neurology and psychiatry department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Autonomics in NMO and MS
Record Dates: First submitted 2025-10-01; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: NMO and MS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bedside cardiovascular reflex tests — These tests evaluate both parasympathetic and sympathetic components of cardiovascular regulation.

SUMMARY:
To compare the frequency and patterns of autonomic dysfunction in patients with NMOSD and MS, and to investigate its correlations with clinical disability, radiological findings, fatigue, and quality of life parameters

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years , both sexes.
* Confirmed diagnosis of NMOSD according to the 2015 International Consensus Criteria.
* Confirmed diagnosis of RRMS according to the 2024 McDonald diagnostic criteria.

Exclusion Criteria:

* Comorbidities affecting autonomic function (e.g., diabetes, Parkinsonism).
* Medications known to interfere with autonomic testing.
* Cognitive impairment precluding questionnaire completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of neuromyelitis optica spectrum disorders and multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of autonomic dysfunction in Neuromyelitis Optica Spectrum Disorder | Baseline
  Autonomic dysfunction assessment using COMPASS-31 questionnaire (Arabic validated version) (12):The Composite Autonomic Symptom Score 31 (COMPASS-31) is a validated, self-administered questionnaire derived from the original 169-item Autonomic Symptom Profile. It provides a concise yet comprehensive evaluation of autonomic symptoms across six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor functions. The total weighted score ranges from 0-100, with higher scores reflecting greater autonomic symptom burden.

SECONDARY OUTCOMES:
Correlations with disability, MRI findings, fatigue, and quality of life. | baseline
  D. Fatigue and psychiatric symptoms
  * Fatigue Severity Scale (FSS): Nine-item scale measuring the impact of fatigue on physical, occupational, and social functioning. Widely validated in MS and NMOSD cohorts.
  * Hamilton Depression Rating Scale (HAM-D)&Hamilton Anxiety Rating Scale (HAM-A): Clinician-administered tools that quantify depression and anxiety severity, respectively. Inclusion is important given the known bidirectional relationship between autonomic dysfunction and mood disorders.
  E. Quality of life. o The SF-36 is a generic health-related quality of life tool with 36 items covering eight domains (physical functioning, role limitations due to physical/emotional health, pain, vitality, mental health, social functioning, and general health).
  A. Neuroimaging: Brain and Spinal MRI
  o MRI will be reviewed for lesion load (number and volume) and lesion topography (anatomical distribution).
  Assessments will be performed by a neuroradiologist blinded to clinical

REFERENCES:
- [Result] BLEWETT J. Manifestations of yaws in Great Britain. Br J Radiol. 1959 Mar;32(375):198-201. doi: 10.1259/0007-1285-32-375-198. No abstract available. PMID 13638541
- [Result] HAMILTON JE, HALL WM, HARBRECHT PJ. Carcinoma of the tongue: its behavior and management. Surgery. 1960 Aug;48:385-90. No abstract available. PMID 14399265
- [Result] Pigg S, Cautley D, Francisco PW. Impacts of weatherization on indoor air quality: A field study of 514 homes. Indoor Air. 2018 Mar;28(2):307-317. doi: 10.1111/ina.12438. Epub 2017 Nov 27. PMID 29108089
- [Result] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Result] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Result] Cohen JA. 2024 revision of the McDonald diagnostic criteria for MS: Substantial and substantive changes. Mult Scler. 2025 Oct;31(11):1269-1275. doi: 10.1177/13524585251351860. Epub 2025 Jul 13. No abstract available. PMID 40652383
- [Result] Pentland B, Ewing DJ. Cardiovascular reflexes in multiple sclerosis. Eur Neurol. 1987;26(1):46-50. doi: 10.1159/000116311. PMID 3816885
- [Result] Wingerchuk DM, Banwell B, Bennett JL, Cabre P, Carroll W, Chitnis T, de Seze J, Fujihara K, Greenberg B, Jacob A, Jarius S, Lana-Peixoto M, Levy M, Simon JH, Tenembaum S, Traboulsee AL, Waters P, Wellik KE, Weinshenker BG; International Panel for NMO Diagnosis. International consensus diagnostic criteria for neuromyelitis optica spectrum disorders. Neurology. 2015 Jul 14;85(2):177-89. doi: 10.1212/WNL.0000000000001729. Epub 2015 Jun 19. PMID 26092914
- [Result] Frileck S. The work. Plast Reconstr Surg. 2003 Aug;112(2):681-3. doi: 10.1097/01.PRS.0000070942.73903.FD. No abstract available. PMID 12900633
- [Result] Crnosija L, Krbot Skoric M, Andabaka M, Junakovic A, Martinovic V, Ivanovic J, Mesaros S, Pekmezovic T, Drulovic J, Habek M. Autonomic dysfunction in people with neuromyelitis optica spectrum disorders. Mult Scler. 2020 May;26(6):688-695. doi: 10.1177/1352458519837703. Epub 2019 Mar 19. PMID 30887872
- [Result] Racosta JM, Kimpinski K. Autonomic dysfunction, immune regulation, and multiple sclerosis. Clin Auton Res. 2016 Feb;26(1):23-31. doi: 10.1007/s10286-015-0325-7. Epub 2015 Dec 21. PMID 26691635
- [Result] Cortez MM, Nagi Reddy SK, Goodman B, Carter JL, Wingerchuk DM. Autonomic symptom burden is associated with MS-related fatigue and quality of life. Mult Scler Relat Disord. 2015 May;4(3):258-63. doi: 10.1016/j.msard.2015.03.007. Epub 2015 Apr 8. PMID 26008943
- [Result] Habek M, Crnosija L, Lovric M, Junakovic A, Krbot Skoric M, Adamec I. Sympathetic cardiovascular and sudomotor functions are frequently affected in early multiple sclerosis. Clin Auton Res. 2016 Dec;26(6):385-393. doi: 10.1007/s10286-016-0370-x. Epub 2016 Jul 22. PMID 27448576
- [Result] Jarius S, Wildemann B. The history of neuromyelitis optica. J Neuroinflammation. 2013 Jan 15;10:8. doi: 10.1186/1742-2094-10-8. PMID 23320783
- [Result] Noyes K, Weinstock-Guttman B. Impact of diagnosis and early treatment on the course of multiple sclerosis. Am J Manag Care. 2013 Nov;19(17 Suppl):s321-31. PMID 24494633